CLINICAL TRIAL: NCT00074750
Title: A Phase I Study of DT388GMCSF Fusion Protein in Acute Myelogenous Leukemia (AML) and Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Study of DT388GMCSF Fusion Protein in Acute Myelogenous Leukemia (AML) and Chronic Myelomonocytic Leukemia (CMML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM03-0130
Record Dates: First submitted 2003-12-19; First posted 2003-12-23 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Acute Myelogenous Leukemia; Chronic Myelomonocytic Leukemia
Keywords: AML; CMML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DTGM (Experimental): Starting dose of DTGM fusion protein 2 mcg/kg/day as a short (30 min) intravenous infusion, three times /week (M,W,F) for two consecutive weeks. In absence of defined grade 3/4 nonhematological toxicities in the first 0/3 or 1/6 patients, the dose will be escalated by 1 mcg/kg/day for the next patient cohort.
  Interventions: Drug: DTGM

INTERVENTIONS:
Drug: DTGM — Starting dose: 2 mcg/kg by vein three times a week (M,W,F) for two consecutive weeks.
  Other Names: Diphtheria toxin fused with granulocyte macrophage colony stimulating factor

SUMMARY:
DTGM belongs to a new generation of drugs designed to target leukemic cells. To achieve this, DTGM takes advantage of the ability of naturally-produced growth factor (GM, granulocyte-macrophage stimulating factor) to deliver a drug (diphtheria toxin) to cells; preferably leukemic cells. It then attaches to the cells and allows the toxin to enter the leukemic cells and destroy them.

DETAILED DESCRIPTION:
The majority of malignant myeloid progenitor cells express receptors for GM-CSF. The fusion of GM-CSF with diphtheria toxin allows a targeting of cells with GM-CSF receptors for effects of the toxin while sparing GM-CSF receptor-lacking multipotent stem cells. The great majority of AML cells express GM-CSF receptors and DT388GMCSF has shown selective killing of AML and CMML progenitors in vitro while sparing normal progenitor cells. When administered as a single bolus to rodents, adequate blood DT388GMCSF biological activity was found to kill several logs of leukemic cells. A phase I clinical trial of DT388GMCSF given as a daily bolus i.v. infusion for up to 5 consecutive days was completed in 38 patients. The study defined liver toxicity as the DLT. The liver toxicity was observed only in patients > 50 years and receiving steroids. Responses were seen in four patients consisting of one complete remission and 3 partial remission of short duration. Peak drug levels were inversely proportional to pre-treatment DT388GMCSF antibody levels.

Because of the observed significant preclinical activity in AML and CMML, clinical activity in chemorefractory patients with AML, the association of toxicities with steroid exposure, and association of the drug level with antibody titer that could be decreased with DT388GMCSF exposure, the current follow up phase I trial is designed based on a new administration and is a dose - finding trial also aimed to better determine and control side effects, improve drug pharmacokinetics and provide initial insight into antileukemic activity of this novel agent, delivered at a prolonged intermittent schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory or relapsed AML ( marrow blasts > 20% ), must have failed induction therapy or have relapsed after CR duration < 6 months following induction therapy, untreated or refractory to salvage chemotherapy. Relapsed AML patients with CR duration > 6 months or previously untreated patients refusing chemotherapy and not considered for treatments of higher priority are also eligible.
* Patients with chronic myelomonocytic leukemia (CMML) who failed at least one course of chemo- or biological therapy( including trial of erythropoietin), or patients with relapsed CMML. Previously untreated CMML patients with HB < or = 12 g / dL, not eligible for protocols of higher priority or not wishing to receive chemotherapy.
* Patients must have an ECOG performance status of < 2.
* Patients must have WBC count < 10,000/mL prior to initiating the treatment. The WBC count must be stabilized below this level for at least three days by leukopheresis or hydroxyurea. Hydroxyurea must be discontinued one day prior to initiation of DT388GMCSF treatment.
* Patients must have creatinine < 1.6 times ULN: bilirubin <1.6 times ULN; SGPT < 2.6 x ULN; albumin > 3 gm/dl; adequate cardiac function (EF >44%), oxygen saturation > 92% without exogenous oxygen administered.
* Patients must be willing to be treated at M D Anderson Cancer Center.
* Women of childbearing potential and men must agree to practice contraception using approved methods.
* No chemotherapy except Hydroxyurea 2 weeks prior to entering the study and recovered from previous toxicity.
* Patients must be > 17 years old.

Exclusion Criteria:

* Patients with serious concurrent medical problems. Patients with proven bacterial infections are not eligible until the resolution of the infection (patient afebrile who completed antibacterial therapy, not on steroids). Patients with active fungal infections are eligible only if evidence of response to antifungal medications is documented and fever does not exceed 38C for at least 2 days.
* Inability to give informed consent because of psychiatric problems or other serious medical problems.
* Pregnant or nursing women.
* Patients with documented CNS leukemia or leukemia with CNS symptoms.
* Patients who have had a myocardial infarction within the past six months.
* Patients with severe penicillin allergy (anaphylaxis).
* Not fully recovered from toxic effects of prior chemotherapy or radiation therapy.
* Patients who are on corticosteroid treatment for any medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miloslav Beran, MD, PhD, DVM, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center's website — http://www.mdanderson.org